CLINICAL TRIAL: NCT02590185
Title: Xploring Venlafaxine Pharmacokinetic Variability by a Phenotyping Approach
Brief Title: MetAbolism vaRiability of VEnLafaxine
Acronym: MARVEL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AOM14562
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Major Depressive Disorders
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cocktail probe drugs (Experimental): * A capsule of omeprazole ABBOTT® 10mg
  * 10 mg of an oral liquid formulation of Dextrométhorphane bromhydrate (Drill Pierre FABRE MEDICAMENT® 5mg/5mL, syrup)
  * 1 mg of an injectable solution of Midazolam for oral administration (Midazolam Panpharma® 1mg/mL, injectable solution)
  * A tablet of fexofenadine Zentiva® 120mg
  Interventions: Drug: cocktail probe drugs

INTERVENTIONS:
Drug: cocktail probe drugs — For the assessment of drug-metabolizing enzyme activity, the patients will be given the cocktail probe drugs, by oral route, one time during the study:
  * A capsule of omeprazole ABBOTT® 10mg
  * 10 mg of an oral liquid formulation of Dextrométhorphane bromhydrate (Drill Pierre FABRE MEDICAMENT® 5mg/5mL, syrup)
  * 1 mg of an injectable solution of Midazolam for oral administration (Midazolam Panpharma® 1mg/mL, injectable solution)
  * A tablet of fexofenadine Zentiva® 120mg

SUMMARY:
Regarding the direct costs and the social value of depression, the decision of an antidepressant treatment prescription must be optimized as much as possible. The development of a personalized medicine in psychiatry may reduce treatment failure, intolerance or resistance, and hence burden and costs of affective disorders.

There is hope that biomarkers will be found to guide treatment selection. It might be of decisive interest to be able to assess an individual's metabolism activity. We propose here to explore the relationship between the activity of drug-metabolizing enzymes (DME) and transporters- assessed by a phenotypic approach and the efficacy of antidepressants. We will focus on venlafaxine (V) that provides a reasonable second-step choice for patients with depression and is used extensively in psychiatric practice, and the metabolism of which involves several cytochromes (CYP) P450 enzymes and the transporter P-gp.

Thus, the primary objective of this study is to study the correlation between the concentration of V and its metabolite ODesmethylV (V+ODV) and drug metabolism variability assessed by a phenotypic approach, in patients with major depressive disorder and MADRS ≥ 20 despite 4 weeks of V at 150mg or less

ELIGIBILITY:
Inclusion Criteria:

* Patient (Hospitalized or outpatient) with major depressive disorder and MADRS ≥ 20 at visit of selection
* Patients non responders to V after 4 weeks of V at 150mg or less
* Decision of the psychiatrist to increase the dose of V at visit of selection
* Understanding of French language and able to give a written inform consent.
* Informed consent signed to participate to the study
* Individuals covered by social security regimen

Exclusion Criteria:

* Patients treated by more than one antidepressant
* Patients currently treated with one of the drug substrate of the cocktail
* Sensitivity or contra-indication to any of the substrate drugs used
* Current pregnancy, desire to get pregnant, or breastfeeding
* Bipolar disorder and schizophrenia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Estimated)
Dates: Start 2015-12; Primary Completion 2019-12 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
The CYP2C19 activity | 2 hours
  5-hydroxyomeprazole/omeprazole
The CYP2D6 activity | 2 hours
  dextrorphan/dextromethorphan ratio
The CYP3A4 activity | 2 hours
  1-hydroxymidazolam/ midazolam ratio
The P-gp activity | 2, 3 and 6 hours
  Fexofenadine AUC based on fexofenadine concentrations

SECONDARY OUTCOMES:
Tobacco use | 20, 40, 70 days
  Fagerstrom test
Mood disorder | 20, 40, 70 days
Anxiety scale Tyrer | 20, 40, 70 days
QIDS-SR16 | 20, 40, 70 days
Criteria for rating medication trials for antidepressant failure and level of resistance | 20, 40, 70 days
MARS Score | 20, 40, 70 days
PRISE-M score | 20, 40, 70 days
FISBER score | 20, 40, 70 days

CONTACTS AND LOCATIONS:
Overall Officials: Celia Lloret-Linares, MD, Principal Investigator — APHP
Locations (2):
- France (2):
  - Fernand Widal hospital, Paris
  - Lariboisiere hospital, Paris

REFERENCES:
- [Derived] Lloret-Linares C, Daali Y, Chevret S, Nieto I, Moliere F, Courtet P, Galtier F, Richieri RM, Morange S, Llorca PM, El-Hage W, Desmidt T, Haesebaert F, Vignaud P, Holtzmann J, Cracowski JL, Leboyer M, Yrondi A, Calvas F, Yon L, Le Corvoisier P, Doumy O, Heron K, Montange D, Davani S, Deglon J, Besson M, Desmeules J, Haffen E, Bellivier F. Exploring venlafaxine pharmacokinetic variability with a phenotyping approach, a multicentric french-swiss study (MARVEL study). BMC Pharmacol Toxicol. 2017 Nov 7;18(1):70. doi: 10.1186/s40360-017-0173-2. PMID 29115994